CLINICAL TRIAL: NCT01673360
Title: Collection of Long Term Patient Outcomes Data Following Implantation of AMS Surgical Devices
Acronym: CAPTURE
Status: Terminated | Type: Observational
Why Stopped: Sponsor is winding down business operations
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: PR1102
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Female Stress Incontinence; Pelvic Organ Prolapse
Keywords: vaginal repair; urinary slings; POP; SUI; prolapse; incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elevate PC: Subjects implanted with Elevate PC
  Interventions: Device: Elevate PC
- Mini Arc Pro: Subjects implanted with Mini Arc Pro
  Interventions: Device: Mini Arc Pro
- RetroArc: Subjects implanted with RetroArc
  Interventions: Device: RetroArc

INTERVENTIONS:
Device: Elevate PC — List of AMS prolapse products
  Groups: Elevate PC
Device: Mini Arc Pro — List of AMS Urinary Incontinence devices
  Groups: Mini Arc Pro
Device: RetroArc — List of AMS Urinary Incontinence devices
  Groups: RetroArc

SUMMARY:
To monitor post-market performance through evaluation of short and long-term performance via:

* Efficacy
* Safety
* Patient reported outcomes

DETAILED DESCRIPTION:
As this is a post-market registry on market approved devices, there will be no formal hypothesis testing. However, points of evaluation will include:

* Characterize the efficacy of the AMS market approved female pelvic health products using standard of care outcome measures and validated quality of life questionnaires
* Characterize the type, severity, and rate of adverse events related to each AMS market approved female pelvic health product
* Collect concomitant procedural data related to the pelvic floor area

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be considered for inclusion in the registry.

  * Have a signed Informed Consent Form
  * Have a signed HIPAA Authorization Form or equivalent Patient Privacy Form if required outside of the US
  * Is a female at least 18 years of age
  * Is scheduled to receive at least one (1) AMS market approved female pelvic health implantable product.
  * Is able and willing to participate in the registry

Exclusion Criteria:

* Patients will be excluded from the registry if any one of the following criteria is met.

  * Patients are contraindicated to receive the target AMS market approved female pelvic health product per the product's IFU

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients planned to receive at least one (1) target AMS market approved female pelvic health product will be considered for inclusion in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2012-09; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Prolapse Efficacy - POP-Q | annually, upto 5 years
  Prolapse Endpoints:
  • POP-Q measurement
Urinary Incontinence Endpoints | annually upto 5 years
  Urinary Incontinence Endpoints:
  * Cough stress test
  * 1 hour pad weight test
  * Urodynamics

CONTACTS AND LOCATIONS:
Locations (19):
- United States (6):
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Womancare, Winston-Salem, North Carolina
  - Seven Hills Women's Health Centers, Cinncinatti, Ohio
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - Female Pelvic Medicine Institute of Virginia, Richmond, Virginia
- Canada (2):
  - The Ottawa Hospital - Shirley E. Greenberg Women's Health Centre, Ottawa, Ontario
  - Windsor Research Office, Windsor, Ontario
- France (2):
  - CMC Beau Soleil, Montpellier
  - Hôpital BICÊTRE, Paris
- Germany (2):
  - German Pelvic Floor Center, St. Hedwig Hospital, Berlin
  - Waldburg-Zeil Kliniken Klinik Tettnang, Tettnang
- University Medical Centre Maribor, Maribor, Slovenia
- Pretoria Urology Hospital, Pretoria, South Africa
- Spain (3):
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital Beata María Ana de Jesus, Madrid
  - Hospital Rio Hortega, Valladolid
- United Kingdom (2):
  - Royal Bolton Hospital, Bolton
  - Glasgow - Southern General Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No